CLINICAL TRIAL: NCT04785625
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of a 300-mg Dose of the INL-001 (Bupivacaine Hydrochloride) Implant in Patients Undergoing Abdominoplasty
Brief Title: Efficacy and Safety Study of Postsurgical Analgesia With INL-001 in Abdominoplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innocoll (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INN-CB-024
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Pain, Postoperative; Abdominoplasty
Keywords: Pain; Analgesia; Postoperative; Abdominoplasty; Bupivacaine; Implant; Postsurgical; Safety; Opioid; Tummy tuck; Efficacy; Post-operative; Post-surgical; Surgery; Placebo; Randomized; Double-blind; Phase 3; Nonopioid; Local anesthetic
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia | interventions — Bupivacaine; Drug Implants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- INL-001 (bupivacaine hydrochloride) implant (Experimental): INL-001 (bupivacaine hydrochloride) implant
  Interventions: Combination Product: Bupivacaine Hydrochloride
- Placebo implant (Placebo Comparator): Placebo collagen-matrix implant
  Interventions: Combination Product: Placebo collagen-matrix implant

INTERVENTIONS:
Combination Product: Bupivacaine Hydrochloride — INL-001 (bupivacaine hydrochloride) implant
  Other Names: XARACOLL (bupivacaine hydrochloride) Implant
  Arms: INL-001 (bupivacaine hydrochloride) implant
Combination Product: Placebo collagen-matrix implant — Placebo collagen-matrix implant
  Arms: Placebo implant

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled efficacy and safety study of the INL-001 (bupivacaine HCl) implant, at 300 mg, in patients following abdominoplasty to evaluate postoperative analgesia.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled efficacy and safety study of the INL-001 (bupivacaine HCl) implant, at 300 mg, in patients following abdominoplasty. Patients will undergo abdominoplasty and have INL-001 or placebo implanted intraoperatively.

The study includes a screening period, an inpatient period (preoperative, intraoperative, immediately postoperative) of approximately 4 days and an outpatient follow-up period (up to 30 days after treatment). Efficacy assessments will be made through 72 hours after treatment (after implant placement). Posttreatment safety assessments will be made throughout the study after the informed consent form is signed, and as specifically scheduled through 72 hours posttreatment, on day 7 (telephone), on day 15 (clinic visit), and on day 30 (clinic visit). Unless the investigator determines further hospitalization is necessary, the patient will be discharged on the day occurring 72 hours after surgery Inpatient day 4).

During the screening period, all patients will undergo eligibility and other screening and safety assessments. On the day of surgery, patient eligibility will be reconfirmed before the start of surgery, patients will be randomly assigned to treatment, and adverse events and prior/concomitant medications will be reviewed. Patients will undergo an abdominoplasty conducted under general anesthesia.

Adverse event and concomitant medication information, including use of rescue pain medication, will be collected throughout the study (inpatient and outpatient). Surgical wound healing/grading assessments and assessment for signs and symptoms potentially indicative of systemic bupivacaine toxicity will be made.

After surgery, patient reports of pain intensity using an 11-point numeric pain rating scale (NPRS) will be recorded at multiple time points through 72 hours posttreatment. Patients will be permitted rescue medication (oral and/or intravenous) to manage breakthrough pain when it occurs.

ELIGIBILITY:
Inclusion Criteria

* Has a body mass index of 18-35 kg/m2.
* Must qualify for a planned (nonemergency) abdominoplasty with rectus sheath plication, with an incision that does not extend beyond the umbilicus, to be performed using standard surgical technique under general anesthesia.
* Has the ability and willingness to comply with all study procedures including being domiciled for at least 72 hours after surgery.
* Is willing to use opioid analgesia, if needed.

Exclusion Criteria

* Has a known hypersensitivity to amide-type local anesthetics, fentanyl, morphine, oxycodone, acetaminophen, NSAIDs, or bovine products.
* Is scheduled for other significant concurrent surgical procedures (eg, gastrointestinal resection or additional cosmetic procedures concurrent with abdominoplasty).
* Has used an opioid analgesic on an extended daily basis (≥5 mg oral morphine equivalents per day for 3 or more days a week) within 4 weeks before surgery and/or chronically uses pain medication.
* Has any chronic painful condition (eg, fibromyalgia), as determined by the investigator, that may confound the assessment of pain associated with the abdominoplasty procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
SPI24 | 0 to 24 hours
  Sum of pain intensity (SPI).The time weighted sum of pain intensity from 0 to 24hours (ie, the area under the NRS PI curve from 0 to 24 hours). For the purpose of SPI computation, Pain Intensity at Time 0 (Baseline PI) is set to zero for all patients who have test article implantation. Minimum value would be "0" and Maximum value would be 240. Time-weighted SPI is calculated as the sum of the pain intensities between successive time points (i.e., if SPI24 = ∑[PI x (time t - time t-1)], where "t" represents a given time point,"t-1" represents the previous time point, and time is expressed in hours). This represents the AUC (Area Under the Curve) of the pain intensities when calculated with the trapezoidal rule.

SECONDARY OUTCOMES:
The secondary objective is to assess the safety and tolerability of INL 001 implants after placement | Day 1 through Day 30
  Safety is assessed and measured by frequency and severity of adverse events

OTHER OUTCOMES:
SPI48 | 0 to 48 hours
  Sum of pain intensity (SPI).The time weighted sum of pain intensity from 0 to 48 hours (ie, the area under the NRS PI curve from 0 to 48 hours). For the purpose of SPI computation, Pain Intensity at Time 0 (Baseline PI) is set to zero for all patients who have test article implantation. Minimum value would be "0" and Maximum value would be 480. Time-weighted SPI is calculated as the sum of the pain intensities between successive time points (i.e., if SPI24 = ∑[PI x (time t - time t-1)], where "t" represents a given time point,"t-1" represents the previous time point, and time is expressed in hours). This represents the AUC (Area Under the Curve) of the pain intensities when calculated with the trapezoidal rule.
SPI72 | 0 to 72 hours
  Sum of pain intensity (SPI). The time weighted sum of pain intensity from 0 to 72 hours (ie, the area under the NRS PI curve from 0 to 72 hours). For the purpose of SPI computation, PI at Time 0 (Baseline PI) is set to zero for all patients who have test article implantation. Where 0 indicates "no pain" and 10 indicated "worst pain possible". A lower score is a better outcome. Minimum value would be "0" and Maximum value would be 720. Time-weighted SPI is calculated as the sum of the pain intensities between successive time points (i.e., if SPI72 = ∑[PI x (time t - time t-1)], where "t" represents a given time point,"t-1" represents the previous time point, and time is expressed in hours). This represents the AUC (Area Under the Curve) of the pain intensities when calculated with the trapezoidal rule.
Proportion of patients who are opioid free through 24 hours | Time 0 through 24 hours
  Proportion of patients who are opioid free through 24 hours
Proportion of patients who are opioid free through 48 hours | Time 0 through 48 hours
  Proportion of patients who are opioid free through 48 hours
Proportion of patients who are opioid free through 72 hours | Time 0 through 72 hours
  Proportion of patients who are opioid free through 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anne Arriaga, Study Director — Lotus Clinical Research
Locations (4):
- United States (4):
  - Lotus Clinical Research, Pasadena, California
  - Midwest Clinical Research, Dayton, Ohio
  - HD Research, Bellaire, Texas
  - Endeavor Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beaton AC, Solanki D, Salazar H, Folkerth S, Singla N, Minkowitz HS, Leiman D, Vaughn B, Skuban N, Niebler G. A randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of a bupivacaine hydrochloride implant in patients undergoing abdominoplasty. Reg Anesth Pain Med. 2023 Dec;48(12):601-607. doi: 10.1136/rapm-2022-104110. Epub 2023 Apr 19. PMID 37076252